CLINICAL TRIAL: NCT00369356
Title: Clinical and Angiographic Outcome of Patients Treated With Bare Metal Stent (BMS) Implantation Compared With Drug Eluting Stents or BMS Plus Systemic Prednisone Therapy. A Randomized, Multicentre Study.
Brief Title: Cortisone or Drug Eluting Stents (DES) as Compared to Bare Metal Stents (BMS) to EliminAte Restenosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Regione Piemonte (Other)
Responsible Party: Principal Investigator, Flavio Ribichini, MD, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEREA-DES
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Sham Comparator): Bare Metal Stenting
  Interventions: Device: Bare metal coronary stent
- 2 (Active Comparator): Stenting with DES
  Interventions: Device: Drug eluting coronary stent
- 3 (Experimental): Bare metal stenting and administration of prednisone
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Bare metal stenting with administration of oral prednisone as described in the protocol
  Arms: 3
Device: Drug eluting coronary stent — Stenting with DES (Cypher or Taxus)
  Arms: 2
Device: Bare metal coronary stent — Stenting with BMS only
  Arms: 1

SUMMARY:
The possibility of using the new drug eluting stents (DES) technology has significantly changed the mid-term outcome of percutaneous coronary interventions (PCI) in terms of reduced recurrence of angina. The way interventionalists accomplish their work is changing accordingly, with a strong trend to a wider use of DES and a consequent perceived patients' clinical benefit.

Evidences supporting the superiority of DES in reducing ischemic recurrence after PCI compared to traditional stents (BMS) are available from randomized studies. A recent meta-analyses underlines that:

DES are superior to BMS in reducing clinical recurrence of ischemia, DES and BMS offer identical results in terms of death and infarction, Rapamycin and paclitaxel DES offer similar results.

The aim of our study is to perform a multicenter, randomized study to assess the clinical efficacy and safety of the oral prednisone therapy after PCI as a possible systemic alternative to currently available BMS and DES. Furthermore, the study aims at analyzing the clinical outcome of the commercially available DES in the context of an independent research and a cost-benefit comparison with BMS and oral steroids.

DETAILED DESCRIPTION:
Design of the study

It is very important to underline that this is a "spontaneous" study, i.e. not receiving sponsorship from pharmaceutical industries, stent manufacturers, or any other financial source. This independence from economic interests would contribute to exclude conflicts of interest that may bias the results of the study that is aimed at testing the applicability and the clinical efficacy of this therapy. Furthermore, the assessment of the DES in public hospitals, and beyond the spectrum of the industry-supported studies may offer interesting results of the real life use of these devices.

One of the purposes of the study is a cost-effectiveness analysis. Centers participating in the study should therefore perform PCI according to their common practice with no interference in their decision-making process or technical approach to PCI because of the inclusion of the patients into a randomized study; this is aimed at obtaining an as real as possible situation of the daily practice. Being an spontaneous research, neither a fee will be provided for the enrollment of patients, nor free stents will be given.

The allocation of patients into a BMS or DES treatment will be decided by randomization, and the stents implanted will be selected according to the operator's preference.

The study will include three different groups of patients:

* Control group: receiving BMS;
* DES group: receiving DES;
* Prednisone group: receiving BMS and oral prednisone

Principal objective of the study: is the comparison of the primary endpoint obtained in a control group of patients treated with BMS versus two alternative study groups:

* DES
* BMS and oral prednisone All assuming a similar adjunctive conventional medical treatment.

Secondary endpoint of the study are:

* cost-effectiveness analysis. This will be calculated considering all patients enrolled in the study and analyzed after one year of the treatment. The analysis will take into account the procedural cost of the PCI material, the cost of the medical treatment in the first year of follow-up and the number of event-free days at follow-up. The cost-efficacy analysis will be obtained from the ratio between the cost of the event-free day of follow-up and the possibility of MACE considered in the primary endpoint of the study.
* comparison of the angiographic results. This will be calculated in all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed CAD (either SVD or MVD) with signs or symptoms of myocardial ischemia, scheduled for percutaneous revascularization are all candidates.
* Either native vessels and SVG can be included with de-novo or recurrent lesions.
* Lesions causing a diameter stenosis >50% in a main coronary artery (LAD, RCA, LCx) or their principal branches (Dg, OM, PL, PDA).

Exclusion Criteria:

* Diabetes
* Age over 80 years old
* Recent Q wave myocardial infarction (less than 2 weeks)
* Severe hypertension, uncontrolled despite medical treatment
* Gastric ulcer or symptomatic gastritis
* Neoplasia
* Renal failure (creatinine >2.5)
* Left main disease, or left main equivalent (proximal LAD and proximal LCx), or three vessel disease involving the proximal segments of the 3 main coronary branches
* Suboptimal angiographic result of PCI (DS% >30% or TIMI flow <grade 3)
* Contraindications to high-doses of steroids (immunosuppression, active infective disease, osteoporosis, recent use of high doses of steroids).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac death, myocardial infarction, recurrence of angina at rest or need to repeat revascularization at 12 months. | 12 months

SECONDARY OUTCOMES:
Angiographic restenosis according to the late loss measurement after 6 to 9 months of the procedure. A DS% =>50 at in-segment analysis will be considered as restenosis. | 9 months
Cost-efficacy analysis of the study at 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Vassanelli, MD, Study Chair — Università di Verona; Flavio Ribichini, MD, Study Director — Università di Verona; Valeria Ferrero, MD, Principal Investigator — Università di Verona
Locations (5):
- Italy (5):
  - Istituto Clinico Humanitas, Milan, Milano
  - Ospedale Maggiore della Carità, Novara, Novara
  - European Hospital, Rome, Rome
  - Ospedale San Giovanni Bosco, Torino, Torino
  - Università di Verona, Verona, Verona

REFERENCES:
- [Background] Versaci F, Gaspardone A, Tomai F, Ribichini F, Russo P, Proietti I, Ghini AS, Ferrero V, Chiariello L, Gioffre PA, Romeo F, Crea F; Immunosuppressive Therapy for the Prevention of Restenosis after Coronary Artery Stent Implantation Study. Immunosuppressive Therapy for the Prevention of Restenosis after Coronary Artery Stent Implantation (IMPRESS Study). J Am Coll Cardiol. 2002 Dec 4;40(11):1935-42. doi: 10.1016/s0735-1097(02)02562-7. PMID 12475452
- [Background] Ribichini F, Ferrero V, Agostini M, Vassanelli C. Immunosuppression against restenosis. Efficacy of a radiofrequency guidewire and oral prednisone in achieving and maintaining coronary artery patency after stenting. Cardiovasc Revasc Med. 2005 Jul-Sep;6(3):124-5. doi: 10.1016/j.carrev.2005.08.006. No abstract available. PMID 16275609
- [Background] Ferrero V, Ribichini F, Rognoni A, Marino P, Brunelleschi S, Vassanelli C. Comparison of efficacy and safety of lower-dose to higher-dose oral prednisone after percutaneous coronary interventions (the IMPRESS-LD study). Am J Cardiol. 2007 Apr 15;99(8):1082-6. doi: 10.1016/j.amjcard.2006.11.064. Epub 2007 Mar 6. PMID 17437731
- [Background] Ribichini F, Ferrero V, Rognoni A, Marino P, Brunelleschi S, Vassanelli C. Percutaneous treatment of coronary bifurcations: lesion preparation before provisional bare metal stenting and subsequent immunosuppression with oral prednisone. The IMPRESS-Y study. J Interv Cardiol. 2007 Apr;20(2):114-21. doi: 10.1111/j.1540-8183.2007.00250.x. PMID 17391219
- [Background] Ribichini F, Tomai F, Paloscia L, Di Sciascio G, Carosio G, Romano M, Verna E, Galli M, Tamburino C, De Cesare N, Pirisi R, Piscione F, Lanteri G, Ferrero V, Vassanelli C; DESIRE investigators. Steroid-eluting stents in patients with acute coronary syndrome: the dexamethasone eluting stent Italian registry. Heart. 2007 May;93(5):598-600. doi: 10.1136/hrt.2006.098467. Epub 2006 Sep 27. PMID 17005712
- [Background] Ribichini F, Joner M, Ferrero V, Finn AV, Crimins J, Nakazawa G, Acampado E, Kolodgie FD, Vassanelli C, Virmani R. Effects of oral prednisone after stenting in a rabbit model of established atherosclerosis. J Am Coll Cardiol. 2007 Jul 10;50(2):176-85. doi: 10.1016/j.jacc.2007.03.031. Epub 2007 Jun 22. PMID 17616304
- [Background] Ferrero V, Ribichini F, Pesarini G, Brunelleschi S, Vassanelli C. Glucocorticoids in the prevention of restenosis after coronary angioplasty: therapeutic potential. Drugs. 2007;67(9):1243-55. doi: 10.2165/00003495-200767090-00001. PMID 17547469
- [Result] Ribichini F, Tomai F, De Luca G, Boccuzzi G, Presbitero P, Pesarini G, Ferrero V, Ghini AS, Abukaresh R, Aurigemma C, De Luca L, Zavalloni D, Soregaroli D, Marino P, Garbo R, Zanolla L, Vassanelli C; CEREA-DES investigators. Immunosuppressive therapy with oral prednisone to prevent restenosis after PCI. A multicenter randomized trial. Am J Med. 2011 May;124(5):434-43. doi: 10.1016/j.amjmed.2010.11.027. PMID 21531233
- [Derived] Ribichini F, Tomai F, Pesarini G, Zivelonghi C, Rognoni A, De Luca G, Boccuzzi G, Presbitero P, Ferrero V, Ghini AS, Marino P, Vassanelli C; CEREA-DES Investigators. Long-term clinical follow-up of the multicentre, randomized study to test immunosuppressive therapy with oral prednisone for the prevention of restenosis after percutaneous coronary interventions: Cortisone plus BMS or DES veRsus BMS alone to EliminAte Restenosis (CEREA-DES). Eur Heart J. 2013 Jun;34(23):1740-8. doi: 10.1093/eurheartj/eht079. Epub 2013 Mar 14. PMID 23492671
- [Derived] Ribichini F, Tomai F, De Luca G, Boccuzzi G, Presbitero P, Pesarini G, Ferrero V, Ghini AS, Pastori F, De Luca L, Zavalloni D, Soregaroli D, Garbo R, Franchi E, Marino P, Minelli M, Vassanelli C. A multicenter, randomized study to test immunosuppressive therapy with oral prednisone for the prevention of restenosis after percutaneous coronary interventions: cortisone plus BMS or DES versus BMS alone to eliminate restenosis (CEREA-DES) - study design and rationale. J Cardiovasc Med (Hagerstown). 2009 Feb;10(2):192-9. doi: 10.2459/JCM.0b013e32831f9176. PMID 19377384
- See also: website containing detailed protocol and info for the patient and the GP (needs registration). Contains also the web-based CRF (only available for participating centers) — http://www.cuorediverona.it